CLINICAL TRIAL: NCT05554302
Title: Characterization of 18F-Fluciclovine PET Amino Acid Radiotracer in Resected Brain Metastasis
Acronym: CONCORDANT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-KOT-003
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Brain Metastases; Brain Cancer
Keywords: Brain metastases; Brain cancer; Stereotactic radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PET/CT, MRI (Experimental): All patients will obtain an 18F-Fluciclovine PET/CT scan in addition to the planning MRI at the time of SRS treatment (approximately 2-4 weeks after resection). The value of 18F-Fluciclovine in addition to structural information from the MRI will be analyzed. Patients will continue to undergo 18F-Fluciclovine in addition to MRI during routine follow-up to determine the ability of 18F-Fluciclovine PET/CT to identify areas at risk for marginal failure, monitor resection beds for tumor control, identify patients at risk for disease recurrence, and detect patterns of failure.
  Interventions: Drug: 18F-Fluciclovine

INTERVENTIONS:
Drug: 18F-Fluciclovine — Patients will receive 5-mCi dose (+/- 20%) of 18F-Fluciclovine intravenously as a bolus injection. They will be required to fast for at least four hours prior to 18F-Fluciclovine injection. Patients will be positioned for PET/CT brain imaging and will be injected with 18F-Fluciclovine immediately prior to PET data acquisition. PET data will be collected in list mode up to 25 minutes post-injection. PET images will be reconstructed in two ways: as a standard static image of data acquired between 10 to 20 minutes post-injection, and as a dynamic series of four 5-minute frames between 5 to 25 minutes post-injection to allow for motion assessment and correction and time-dependent observations.

SUMMARY:
This study is for patients who have had surgery to remove brain metastasis and are planned to have stereotactic radiosurgery (SRS) after their brain surgery. It will be optional for patients to have a pre-surgery 18F-Fluciclovine PET/CT scan. The goal of the study is to determine whether a specific imaging agent, known as 18F-Fluciclovine, will help physicians evaluate the extent of surgery and determine if there is any visible tumor above what MRI alone can identify as well as improve the physicians' ability to detect recurring disease. This agent (18F-Fluciclovine) is investigational for the imaging of brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Performance status, Eastern Cooperative Oncology Group (ECOG) 0-3
3. Radiographic diagnosis of brain metastasis
4. Patient planned for surgical intervention for at least 1 metastasis
5. Patient planned for postoperative SRS

Male or female patients of reproductive potential need to employ two highly effective and acceptable forms of contraception for at least 4 weeks prior to screening and agreement to use such a method during study participation and for an additional 1 week after post-treatment 18F-Fluciclovine PET/CT. Highly effective and acceptable forms of contraception are:

* Male condom plus spermicide
* Cap plus spermicide
* Diaphragm plus spermicide
* Copper T
* Progesterone T
* Levonorgestrel-releasing intrauterine system (e.g., Mirena®)
* Implants
* Hormone shot or injection
* Combined pill
* Mini-pill
* Patch

Postmenopausal people on the study (that will not need contraception) is defined as at least one of the following:

* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50
* Radiation-induced oophorectomy with last menses > 1 year ago
* Chemotherapy-induced menopause with >1 year interval since last menses
* Surgical sterilization (bilateral oophorectomy or hysterectomy).

Exclusion Criteria:

1. Prior anaphylactic reaction to 18F-Fluciclovine
2. Evidence of leptomeningeal disease
3. Prior whole-brain radiation therapy
4. Contraindication to MRI (e.g., due to safety reasons, such as presence of a pacemaker)
5. Pregnant at the expected time of 18F-fluciclovine administration
6. Expecting to be breastfeeding at the time of 18F-Fluciclovine and unwilling to stop breast-feeding for 24 hours. Temporary cessation of breastfeeding 24 hours after the time of imaging is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change in conformality index of tumor target volume delineation | 3 weeks, 6 and 12 months
  The tumor target volume (post-operative cavity and any residual or recurrent disease) will be delineated by post-operative MRI only. A second target volume will be generated using the 18F-Fluciclovine PET-defined volume. The conformality index is calculated by comparing the PET-defined tumor volume with MRI-defined tumor volume. Non-overlapping and overlapping regions regions of PET tumor volume and MRI tumor volume will be used to calculate conformality indices.
Change in PET scan standardized uptake value (SUV) parameters | 3 weeks, 6 and 12 months
  The standardized uptake value (SUV) parameters of SUVpeak, SUVmean, and SUVmax will be measured to determine if they correlate tumor volume and can predict risk of recurrence.

SECONDARY OUTCOMES:
Time to local failure | 1 year
  Each lesion will be followed from pre-treatment PET to local failure or re-retreatment; death; 12 months from pre-treatment PET; lost-to follow-up, discontinuation, or withdrawal; or end of study. In the event that a patient has more than one study eligible lesion, the patient will discontinue follow up after all lesions progress, or will be censored as above. Death will be treated as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh R Kotecha, M.D., Principal Investigator — Miami Cancer Institute/Baptist Health South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kotecha R, Gondi V, Ahluwalia MS, Brastianos PK, Mehta MP. Recent advances in managing brain metastasis. F1000Res. 2018 Nov 9;7:F1000 Faculty Rev-1772. doi: 10.12688/f1000research.15903.1. eCollection 2018. PMID 30473769
- [Background] Kotecha R, Ahluwalia MS, Siomin V, McDermott MW. Surgery, Stereotactic Radiosurgery, and Systemic Therapy in the Management of Operable Brain Metastasis. Neurol Clin. 2022 May;40(2):421-436. doi: 10.1016/j.ncl.2021.11.002. Epub 2022 Mar 31. PMID 35465884
- [Background] Soltys JS, Wilson SE. Directional sensitivity of velocity sense in the lumbar spine. J Appl Biomech. 2008 Aug;24(3):244-51. doi: 10.1123/jab.24.3.244. PMID 18843154
- [Background] Choi HJ, Choi SK, Lim YJ. Radiosurgical techniques and clinical outcomes of gamma knife radiosurgery for brainstem arteriovenous malformations. J Korean Neurosurg Soc. 2012 Dec;52(6):534-40. doi: 10.3340/jkns.2012.52.6.534. Epub 2012 Dec 31. PMID 23346325
- [Background] Jhaveri J, Chowdhary M, Zhang X, Press RH, Switchenko JM, Ferris MJ, Morgan TM, Roper J, Dhabaan A, Elder E, Eaton BR, Olson JJ, Curran WJ, Shu HG, Crocker IR, Patel KR. Does size matter? Investigating the optimal planning target volume margin for postoperative stereotactic radiosurgery to resected brain metastases. J Neurosurg. 2019 Mar 1;130(3):797-803. doi: 10.3171/2017.9.JNS171735. Epub 2018 Apr 20. PMID 29676690
- [Background] Gui C, Moore J, Grimm J, Kleinberg L, McNutt T, Shen C, Chen L, Bettegowda C, Lim M, Redmond KJ. Local recurrence patterns after postoperative stereotactic radiation surgery to resected brain metastases: A quantitative analysis to guide target delineation. Pract Radiat Oncol. 2018 Nov-Dec;8(6):388-396. doi: 10.1016/j.prro.2018.04.010. Epub 2018 Apr 26. PMID 30029965
- [Background] Shi S, Sandhu N, Jin M, Wang E, Liu E, Jaoude JA, Schofield K, Zhang C, Gibbs IC, Hancock SL, Chang SD, Li G, Gephart MH, Pollom EL, Soltys SG. Stereotactic Radiosurgery for Resected Brain Metastases: Does the Surgical Corridor Need to be Targeted? Pract Radiat Oncol. 2020 Sep-Oct;10(5):e363-e371. doi: 10.1016/j.prro.2020.04.009. Epub 2020 May 16. PMID 32428766
- [Background] Soliman H, Ruschin M, Angelov L, Brown PD, Chiang VLS, Kirkpatrick JP, Lo SS, Mahajan A, Oh KS, Sheehan JP, Soltys SG, Sahgal A. Consensus Contouring Guidelines for Postoperative Completely Resected Cavity Stereotactic Radiosurgery for Brain Metastases. Int J Radiat Oncol Biol Phys. 2018 Feb 1;100(2):436-442. doi: 10.1016/j.ijrobp.2017.09.047. Epub 2017 Oct 4. PMID 29157748
- [Background] Galldiks N, Langen KJ. Amino acid PET in neuro-oncology: applications in the clinic. Expert Rev Anticancer Ther. 2017 May;17(5):395-397. doi: 10.1080/14737140.2017.1302799. Epub 2017 Mar 11. No abstract available. PMID 28277832
- [Background] Albert NL, Weller M, Suchorska B, Galldiks N, Soffietti R, Kim MM, la Fougere C, Pope W, Law I, Arbizu J, Chamberlain MC, Vogelbaum M, Ellingson BM, Tonn JC. Response Assessment in Neuro-Oncology working group and European Association for Neuro-Oncology recommendations for the clinical use of PET imaging in gliomas. Neuro Oncol. 2016 Sep;18(9):1199-208. doi: 10.1093/neuonc/now058. Epub 2016 Apr 21. PMID 27106405
- [Background] Okudaira H, Shikano N, Nishii R, Miyagi T, Yoshimoto M, Kobayashi M, Ohe K, Nakanishi T, Tamai I, Namiki M, Kawai K. Putative transport mechanism and intracellular fate of trans-1-amino-3-18F-fluorocyclobutanecarboxylic acid in human prostate cancer. J Nucl Med. 2011 May;52(5):822-9. doi: 10.2967/jnumed.110.086074. PMID 21536930
- [Background] Oka S, Okudaira H, Yoshida Y, Schuster DM, Goodman MM, Shirakami Y. Transport mechanisms of trans-1-amino-3-fluoro[1-(14)C]cyclobutanecarboxylic acid in prostate cancer cells. Nucl Med Biol. 2012 Jan;39(1):109-19. doi: 10.1016/j.nucmedbio.2011.06.008. Epub 2011 Sep 29. PMID 21958853
- [Background] Ono M, Oka S, Okudaira H, Schuster DM, Goodman MM, Kawai K, Shirakami Y. Comparative evaluation of transport mechanisms of trans-1-amino-3-[(1)(8)F]fluorocyclobutanecarboxylic acid and L-[methyl-(1)(1)C]methionine in human glioma cell lines. Brain Res. 2013 Oct 16;1535:24-37. doi: 10.1016/j.brainres.2013.08.037. Epub 2013 Aug 27. PMID 23994214
- [Background] Doi Y, Kanagawa M, Maya Y, Tanaka A, Oka S, Nakata N, Toyama M, Matsumoto H, Shirakami Y. Evaluation of trans-1-amino-3-18F-fluorocyclobutanecarboxylic acid accumulation in low-grade glioma in chemically induced rat models: PET and autoradiography compared with morphological images and histopathological findings. Nucl Med Biol. 2015 Aug;42(8):664-72. doi: 10.1016/j.nucmedbio.2015.04.008. Epub 2015 May 7. PMID 26022202
- [Background] Sasajima T, Ono T, Shimada N, Doi Y, Oka S, Kanagawa M, Baden A, Mizoi K. Trans-1-amino-3-18F-fluorocyclobutanecarboxylic acid (anti-18F-FACBC) is a feasible alternative to 11C-methyl-L-methionine and magnetic resonance imaging for monitoring treatment response in gliomas. Nucl Med Biol. 2013 Aug;40(6):808-15. doi: 10.1016/j.nucmedbio.2013.04.007. Epub 2013 May 21. PMID 23701701
- [Background] Oka S, Okudaira H, Ono M, Schuster DM, Goodman MM, Kawai K, Shirakami Y. Differences in transport mechanisms of trans-1-amino-3-[18F]fluorocyclobutanecarboxylic acid in inflammation, prostate cancer, and glioma cells: comparison with L-[methyl-11C]methionine and 2-deoxy-2-[18F]fluoro-D-glucose. Mol Imaging Biol. 2014 Jun;16(3):322-9. doi: 10.1007/s11307-013-0693-0. PMID 24136390
- [Background] Parent EE, Patel D, Nye JA, Li Z, Olson JJ, Schuster DM, Goodman MM. [18F]-Fluciclovine PET discrimination of recurrent intracranial metastatic disease from radiation necrosis. EJNMMI Res. 2020 Dec 7;10(1):148. doi: 10.1186/s13550-020-00739-6. PMID 33284388
- [Background] Kondo A, Ishii H, Aoki S, Suzuki M, Nagasawa H, Kubota K, Minamimoto R, Arakawa A, Tominaga M, Arai H. Phase IIa clinical study of [18F]fluciclovine: efficacy and safety of a new PET tracer for brain tumors. Ann Nucl Med. 2016 Nov;30(9):608-618. doi: 10.1007/s12149-016-1102-y. Epub 2016 Jul 14. PMID 27418267
- [Background] Wakabayashi T, Iuchi T, Tsuyuguchi N, Nishikawa R, Arakawa Y, Sasayama T, Miyake K, Nariai T, Narita Y, Hashimoto N, Okuda O, Matsuda H, Kubota K, Ito K, Nakazato Y, Kubomura K. Diagnostic Performance and Safety of Positron Emission Tomography Using 18F-Fluciclovine in Patients with Clinically Suspected High- or Low-grade Gliomas: A Multicenter Phase IIb Trial. Asia Ocean J Nucl Med Biol. 2017 Winter;5(1):10-21. doi: 10.22038/aojnmb.2016.7869. PMID 28840134
- [Background] Parent EE, Benayoun M, Ibeanu I, Olson JJ, Hadjipanayis CG, Brat DJ, Adhikarla V, Nye J, Schuster DM, Goodman MM. [18F]Fluciclovine PET discrimination between high- and low-grade gliomas. EJNMMI Res. 2018 Jul 25;8(1):67. doi: 10.1186/s13550-018-0415-3. PMID 30046944
- [Background] Tsuyuguchi N, Terakawa Y, Uda T, Nakajo K, Kanemura Y. Diagnosis of Brain Tumors Using Amino Acid Transport PET Imaging with 18F-fluciclovine: A Comparative Study with L-methyl-11C-methionine PET Imaging. Asia Ocean J Nucl Med Biol. 2017 Spring;5(2):85-94. doi: 10.22038/aojnmb.2017.8843. PMID 28660218
- [Background] Wakabayashi T, Hirose Y, Miyake K, Arakawa Y, Kagawa N, Nariai T, Narita Y, Nishikawa R, Tsuyuguchi N, Fukami T, Sasaki H, Sasayama T, Kondo A, Iuchi T, Matsuda H, Kubota K, Minamimoto R, Terauchi T, Nakazato Y, Kubomura K, Wada M. Determining the extent of tumor resection at surgical planning with 18F-fluciclovine PET/CT in patients with suspected glioma: multicenter phase III trials. Ann Nucl Med. 2021 Dec;35(12):1279-1292. doi: 10.1007/s12149-021-01670-z. Epub 2021 Aug 18. PMID 34406623
- [Background] Gondi V, Bradley K, Mehta M, Howard A, Khuntia D, Ritter M, Tome W. Impact of hybrid fluorodeoxyglucose positron-emission tomography/computed tomography on radiotherapy planning in esophageal and non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):187-95. doi: 10.1016/j.ijrobp.2006.09.033. PMID 17189070